CLINICAL TRIAL: NCT02316223
Title: Clinic-based vs. Home-based Support to Improve Care and Outcomes for Older Asthmatics
Brief Title: Supporting Asthma Management Behaviors in Aging Adults
Acronym: SAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 13-1401; AS-1307-05584 (Other: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Asthma
Keywords: asthma; high-risk; adult; elderly; care coordination; community health worker; electronic medical record
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinic-based care coordination (Experimental): The ACC and CHW programs for asthma CC/SMS will have the same objectives and provide the same general services at the office/clinic. The ACC and CHW programs were developed from existing, successfully operating programs at the participating sites, and in the East Harlem and South Bronx communities.
  Interventions: Behavioral: Supporting Asthma Management Behaviors in Aging Adults (SAMBA)
- Home-based care coordination (Active Comparator): The ACC and CHW programs for asthma CC/SMS will have the same objectives and provide the same general services at participant's home. The ACC and CHW programs were developed from existing, successfully operating programs at the participating sites, and in the East Harlem and South Bronx communities.
  Interventions: Behavioral: Supporting Asthma Management Behaviors in Aging Adults (SAMBA)
- Usual care (No Intervention): Clinician-centric strategy and EMR-based clinician decision support

INTERVENTIONS:
Behavioral: Supporting Asthma Management Behaviors in Aging Adults (SAMBA) — The SAMBA program will be led by an asthma care coach (ACC) and the home program by a community health worker (CHW). All interventions, including usual care, will include EMR-based asthma self-management and decision support tools for clinicians in all practice sites. The ACC and CHW will provide education, goal setting, and general self-management support with assigned patients and coordinate with PCPs through in-person and phone contacts over 12 months. Outcomes will be measured through interviews, EMR chart abstractions, and from the Statewide Planning and Research Cooperative System (SPARCS) dataset to identify all ED visits and hospitalizations to any New York State facility.
  Other Names: SAMBA
  Arms: Clinic-based care coordination; Home-based care coordination

SUMMARY:
A 3-arm, patient-randomized trial among Latino and African-American older adults with poorly-controlled asthma will be conducted to compare the effectiveness of clinic-based vs. home-based asthma care coordination / self-management support (CC/SMS) vs. usual care.

DETAILED DESCRIPTION:
Older asthmatics experience worse outcomes than younger adults, especially if they identify as Latino or African-American. Several factors contribute to worse outcomes in these populations including frailty, cognitive impairment, managing multiple chronic diseases and multiple daily medications, low health literacy and English proficiency, high healthcare costs, and misunderstandings about asthma. To our knowledge, there are no programs designed to help older asthmatics manage their illness. In order to address these factors two emerging patient-centered strategies, clinic- and home-based care coordination and self-management support led by an Asthma Care Coach (ACC) and a community health worker (CHW), respectively, will be tested. These strategies will be combined a clinician-centered strategy, use of electronic medical record (EMR)-based asthma decision support that guides medication prescribing, basic counseling, and provision of asthma action plans.

Specific aims are:

1. To compare the effectiveness of (1) ACC/clinic- or (2) CHW/home-based asthma care coordination and self-management support with (3) no care coordination/self-management support (usual care) for improving asthma-related outcomes;
2. To identify subsets of individuals who have greater benefit from home-based care coordination and self-management support compared to clinic-based support.

A 3-arm, randomized trial will be conducted among 450 adult asthmatics ages 60 and older at primary care practices in East and Central Harlem and the South Bronx. All patients, regardless of assignment, will receive care from primary care providers (PCP) with access to the EMR-based asthma decision support. Patients in the ACC and CHW arms will be assessed for barriers to asthma control and will receive support specifically tailored to the identified barriers, including those arising from physical, mental, social/economic, or cognitive issues. Program participation will be 12 months, during which the ACCs and CHWs will also work with the patients' PCPs to optimize care. The study team will engage stakeholders (patients and caregivers, clinicians, community-based organizations, others) to develop and prepare study materials and protocols. In addition to studying patient outcomes, the process of implementing these models of care will be evaluated and documented.

Patients in the ACC and CHW arms will have similar asthma outcomes (asthma control, quality of life, use of urgent care, appointment keeping, medication adherence, use of asthma actions plans). Compared to usual care, patients in the ACC and CHW arms will perform better on these outcomes. Patients with more severe asthma and those at greater risk of missed clinic appointments because of physical or cognitive impairment and psychosocial issues (e.g., substance abuse, mental illness) will be more likely to benefit from the CHW/home-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* ages ≤60 years
* physician diagnosis of asthma
* English- or Spanish-speaking

Exclusion Criteria:

* physician diagnosis of Chronic Obstructive Pulmonary Disease (COPD) or other chronic lung condition
* ≤15 pack-years
* enrollment in another asthma self-management program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2015-01; Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Federman, MD,MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - The Institute for Family Health, New York, New York
  - Mount Sinai-St. Luke's Roosevelt Hospital Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Federman AD, Thanik E, O'Conor R, Arora A, Wolf MS, Wisnivesky JP. Patient characteristics associated with improvements in asthma control and reduction in emergency department visits for older adults with asthma. J Asthma. 2021 Nov;58(11):1528-1535. doi: 10.1080/02770903.2020.1805753. Epub 2020 Aug 19. PMID 32812836
- [Derived] Federman AD, O'Conor R, Mindlis I, Hoy-Rosas J, Hauser D, Lurio J, Shroff N, Lopez R, Erblich J, Wolf MS, Wisnivesky JP. Effect of a Self-management Support Intervention on Asthma Outcomes in Older Adults: The SAMBA Study Randomized Clinical Trial. JAMA Intern Med. 2019 Aug 1;179(8):1113-1121. doi: 10.1001/jamainternmed.2019.1201. PMID 31180474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from 2015 to 2017
Groups:
- Clinic-based Care Coordination: Supporting Asthma Management Behaviors in Aging Adults (SAMBA): The SAMBA program will be led by an asthma care coach (ACC). The ACC will provide education, goal setting, and general self-management support with assigned patients and coordinate with PCPs through in-person and phone contacts over 12 months.
- Home-based Care Coordination: Supporting Asthma Management Behaviors in Aging Adults (SAMBA): The SAMBA program will be led by an asthma care coach (ACC) and the home program by a community health worker (CHW). The ACC and CHW will provide education, goal setting, and general self-management support with assigned patients and coordinate with PCPs through in-person and phone contacts over 12 months.
Period: Overall Study
Arm/Group | Clinic-based Care Coordination | Home-based Care Coordination | Usual Care
Started | 134 | 133 | 139
Completed | 90 | 76 | 95
Not Completed | 44 | 57 | 44
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Lost to Follow-up | 27 | 34 | 36
Not completed — COPD Diagnosis | 3 | 2 | 3
Not completed — Reside outside study area | 1 | 1 | 1
Not completed — No asthma | 2 | 0 | 0
Not completed — Discontinued by PI | 11 | 19 | 3

BASELINE CHARACTERISTICS:
Population: Only those who received the allocated intervention were included in the analysis.
Groups:
- Home-based Care Coordination: Supporting Asthma Management Behaviors in Aging Adults (SAMBA): The SAMBA program will be led by an asthma care coach (ACC) and the home program by a community health worker (CHW). The CHW will provide education, goal setting, and general self-management support with assigned patients and coordinate with PCPs through in-person and phone contacts over 12 months.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Home-based Care Coordination | Clinic-based Care Coordination | Total
Number analyzed (Participants) | 134 | 128 | 129 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.1) | 67.8 (7.4) | 66.5 (6.4) | 67.3 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  60-69 | 88 | 84 | 98 | 270
  70-79 | 27 | 32 | 24 | 83
  80+ | 19 | 12 | 7 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 109 | 107 | 333
  Male | 17 | 19 | 22 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 6 | 12 | 11 | 29
  Black, non-Hispanic | 43 | 37 | 39 | 119
  Hispanic | 76 | 74 | 70 | 220
  Other | 9 | 5 | 9 | 23
Limited English Proficiency [Count of Participants; unit: Participants] | 52 | 49 | 43 | 144
Monthly Household Income <$1350 [Count of Participants; unit: Participants] | 86 | 87 | 89 | 262
Married or Partner [Count of Participants; unit: Participants] | 39 | 33 | 22 | 94
Education Level [Count of Participants; unit: Participants]
  Less than high school | 63 | 50 | 50 | 163
  High school graduate | 27 | 31 | 24 | 82
  Some college | 31 | 25 | 28 | 84
  College graduate | 13 | 22 | 27 | 62
Physical Impairment, severe [Count of Participants; unit: Participants] | 22 | 16 | 20 | 58
Cognitive Impairment [Count of Participants; unit: Participants] | 75 | 63 | 66 | 204
Moderate-severed Depression [Count of Participants; unit: Participants] | 10 | 12 | 10 | 32
Diabetes Mellitus Co-morbid Medical Condition [Count of Participants; unit: Participants] | 52 | 44 | 57 | 153
High Cholesterol Co-morbid Medical Condition [Count of Participants; unit: Participants] | 74 | 70 | 66 | 210
Hypertension Co-morbid Medical Condition [Count of Participants; unit: Participants] | 106 | 88 | 89 | 283

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Test (ACT)
Description: The Asthma Control Test™ is a quick test for people with asthma 12 years and older. The ACT is a 5 items, with 4-week recall (on symptoms and daily functioning) patient self-administered tool for identifying those with poorly controlled asthma. Each items is scored on a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled), The total scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control.
  It provides a numerical score to help assess asthma control at 12 months compared to baseline.
Time Frame: baseline, 3 months, 6 months, and 12 months
Population: only those who completed the respective study visits were included in the data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
Number analyzed (Participants) | 128 | 129 | 134
score on a scale
  Baseline | 15.0 (3.8) | 14.6 (4.0) | 14.3 (4.0)
  3 months | 16.6 (4.4) | 15.7 (4.4) | 14.6 (4.8)
  6 months | 16.8 (4.3) | 15.8 (4.4) | 14.6 (4.9)
  12 months: number analyzed (Participants) | 76 | 90 | 95
  12 months | 17.4 (4.8) | 16.9 (4.7) | 16.1 (4.3)

2. Secondary Outcome: Mini Asthma Quality of Life Questionnaire (AQLQ)
Description: The mini AQLQ is a 15-item self-administered questionnaire, each question scored on a 7-point scale, from 1 (all of the time) to 7 (none of the time) for the first 11 questions, and 1 (totally limited) to 7 (not at all limited) for the last 4 question , with total scale as an average from 1 to 7, with higher score indicating better quality of life or less impairment.
Time Frame: baseline, 3 months, 6 months, and 12 months
Population: only those who completed the respective study visits were included in the data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
Number analyzed (Participants) | 128 | 129 | 134
score on a scale
  Baseline | 4.4 (1.2) | 4.4 (1.2) | 4.3 (1.1)
  3 months | 4.8 (1.8) | 4.6 (1.2) | 4.3 (1.3)
  6 months | 4.9 (1.2) | 4.5 (1.4) | 4.3 (1.3)
  12 months: number analyzed (Participants) | 76 | 90 | 95
  12 months | 4.9 (1.3) | 4.8 (1.4) | 4.6 (1.3)

3. Secondary Outcome: Change in Percent of Patients With >=1 Emergency Dept Visits
Description: Percent of patients with one or more acute asthma-related Emergency Department visits at 12 months compared to baseline for participants in Home-based care coordination and Clinic-based care coordination.
Time Frame: 12 months
Population: only those who completed the study at 12 months were included for the data results for the 12 month mark
Measure: Number; unit: percentage of participants
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
Number analyzed (Participants) | 128 | 129 | 134
percentage of participants
  Baseline | 13.1 | 9.3 | 9.7
  12 months | 7.7 | 6.2 | 12.7

4. Secondary Outcome: Medication Adherence Rating Scale (MARS)
Description: Adherence to ICS and leukotriene receptor antagonists will be assessed with the MARS, a 10-item self-reported measure of adherence to inhaler medications at 12 months compared to baseline. Total scores range from 0 (low likelihood of medication adherence) to 10 (high likelihood), with higher score indicating higher likelihood of medication adherence
Time Frame: baseline, 3 months, 6 months, and 12 months
Population: only those who completed the respective study visits were included in the data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
Number analyzed (Participants) | 128 | 129 | 134
score on a scale
  Baseline | 3.6 (0.7) | 3.7 (0.6) | 3.8 (0.7)
  3 months | 3.9 (0.6) | 3.9 (0.6) | 3.8 (0.7)
  6 months | 3.9 (0.7) | 4.0 (0.7) | 3.8 (0.7)
  12 months: number analyzed (Participants) | 76 | 90 | 95
  12 months | 3.8 (0.8) | 4.0 (0.7) | 3.8 (0.7)

5. Secondary Outcome: Number of Participants With Correct MDI Technique
Description: Number of participants demonstrating MDI technique, correctly completed steps at 12 months as compared to baseline
Time Frame: baseline and 12 months
Population: only those who completed the study at 12 months were included for the data results for the 12 month mark
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
Number analyzed (Participants) | 128 | 129 | 134
Participants
  Baseline | 77 | 71 | 86
  12 months: number analyzed (Participants) | 76 | 90 | 95
  12 months | 54 | 55 | 55

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Home-based Care Coordination | Clinic-based Care Coordination | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/129 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/129 | 0/134
Other Adverse Events (participants affected / at risk) | 0/128 | 0/129 | 0/134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT02316223/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT02316223/SAP_001.pdf